CLINICAL TRIAL: NCT03174899
Title: Role of Diffusion Weighted Magnetic Resonance Imaging in Evaluation of Chronic Kidney Disease
Brief Title: Diffusion Weighted Magnetic Resonance Imaging in Chronic Kidney Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, DMAhmed, Principal investigator, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DMR
Record Dates: First submitted 2017-05-26; First posted 2017-06-05 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Renal Disease
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Stage1:eGFR; ≥90 mL/min/1.73 m2 . (Experimental): All MRI examinations will be performed with a 1.5-T scanner (Acheiva, Philips, and Netherland). All MRI scans will be obtained with the following parameters: Repetition time (TR); 1580 MS, echo time (TE); 60 MS, slice thickness; 1-5 mm, receiver bandwidth; 1158 kHz/pixel, field of view (FOV); 40 cm, matrix size; 164 × 159. . ADC value of the kidneys will be calculated with Diffusion weighted magnetic resonance imaging gradient b-values of 0 and 1000s/mm2. In the axial ADC map, a region of interest (ROI) will be placed for measurement of ADC values on the renal parenchyma of both kidneys, without any preference for cortex or medulla. Three circular ROIs of size 1 cm2 will be placed-one each at the upper pole, inter-polar region, and lower pole of both kidneys-and 6 total ROIs from bilateral kidneys will be averaged for each patient. The mean ADC values will be recorded for each patient and the relationship of ADC values with CKD stage will be evaluated.
  Interventions: Radiation: Diffusion weighted magnetic resonance imaging
- Stage 2: eGFR; 60-89 mL/min/1.73 m2 . (Experimental): All MRI examinations will be performed with a 1.5-T scanner (Acheiva, Philips, and Netherland). All MRI scans will be obtained with the following parameters: Repetition time (TR); 1580 MS, echo time (TE); 60 MS, slice thickness; 1-5 mm, receiver bandwidth; 1158 kHz/pixel, field of view (FOV); 40 cm, matrix size; 164 × 159. ADC value of the kidneys will be calculated with Diffusion weighted magnetic resonance imaging gradient b-values of 0 and 1000s/mm2. In the axial ADC map, a region of interest (ROI) will be placed for measurement of ADC values on the renal parenchyma of both kidneys, without any preference for cortex or medulla. Three circular ROIs of size 1 cm2 will be placed-one each at the upper pole, inter-polar region, and lower pole of both kidneys-and 6 total ROIs from bilateral kidneys will be averaged for each patient. The mean ADC values will be recorded for each patient and the relationship of ADC values with CKD stage will be evaluated.
  Interventions: Radiation: Diffusion weighted magnetic resonance imaging
- Stage 3:eGFR; 30-59 mL/min/1.73 m2 (Experimental): All MRI examinations will be performed with a 1.5-T scanner (Acheiva, Philips, and Netherland). All MRI scans will be obtained with the following parameters: Repetition time (TR); 1580 MS, echo time (TE); 60 MS, slice thickness; 1-5 mm, receiver bandwidth; 1158 kHz/pixel, field of view (FOV); 40 cm, matrix size; 164 × 159. ADC value of the kidneys will be calculated with Diffusion weighted magnetic resonance imaging gradient b-values of 0 and 1000s/mm2. In the axial ADC map, a region of interest (ROI) will be placed for measurement of ADC values on the renal parenchyma of both kidneys, without any preference for cortex or medulla. Three circular ROIs of size 1 cm2 will be placed-one each at the upper pole, inter-polar region, and lower pole of both kidneys-and 6 total ROIs from bilateral kidneys will be averaged for each patient. The mean ADC values will be recorded for each patient and the relationship of ADC values with CKD stage will be evaluated.
  Interventions: Radiation: Diffusion weighted magnetic resonance imaging
- Stage 4:eGFR; 15-29 mL/min/1.73 m2 . (Experimental): All MRI examinations will be performed with a 1.5-T scanner (Acheiva, Philips, and Netherland). All MRI scans will be obtained with the following parameters: Repetition time (TR); 1580 MS, echo time (TE); 60 MS, slice thickness; 1-5 mm, receiver bandwidth; 1158 kHz/pixel, field of view (FOV); 40 cm, matrix size; 164 × 159. ADC value of the kidneys will be calculated with Diffusion weighted magnetic resonance imaginggradient b-values of 0 and 1000s/mm2. In the axial ADC map, a region of interest (ROI) will be placed for measurement of ADC values on the renal parenchyma of both kidneys, without any preference for cortex or medulla. Three circular ROIs of size 1 cm2 will be placed-one each at the upper pole, inter-polar region, and lower pole of both kidneys-and 6 total ROIs from bilateral kidneys will be averaged for each patient. The mean ADC values will be recorded for each patient and the relationship of ADC values with CKD stage will be evaluated.
  Interventions: Radiation: Diffusion weighted magnetic resonance imaging
- Stage 5:eGFR; < 15 mL/min/1.73 m2. (Experimental): All MRI examinations will be performed with a 1.5-T scanner (Acheiva, Philips, and Netherland). All MRI scans will be obtained with the following parameters: Repetition time (TR); 1580 MS, echo time (TE); 60 MS, slice thickness; 1-5 mm, receiver bandwidth; 1158 kHz/pixel, field of view (FOV); 40 cm, matrix size; 164 × 159. ADC value of the kidneys will be calculated with Diffusion weighted magnetic resonance imaging gradient b-values of 0 and 1000s/mm2. In the axial ADC map, a region of interest (ROI) will be placed for measurement of ADC values on the renal parenchyma of both kidneys, without any preference for cortex or medulla. Three circular ROIs of size 1 cm2 will be placed-one each at the upper pole, inter-polar region, and lower pole of both kidneys-and 6 total ROIs from bilateral kidneys will be averaged for each patient. The mean ADC values will be recorded for each patient and the relationship of ADC values with CKD stage will be evaluated.
  Interventions: Radiation: Diffusion weighted magnetic resonance imaging

INTERVENTIONS:
Radiation: Diffusion weighted magnetic resonance imaging — All MRI examinations will be performed with a 1.5-T scanner (Acheiva, Philips, and Netherland). All MRI scans will be obtained with the following parameters: Repetition time (TR); 1580 MS, echo time (TE); 60 MS, slice thickness; 1-5 mm, receiver bandwidth; 1158 kHz/pixel, field of view (FOV); 40 cm, matrix size; 164 × 159. ADC value of the kidneys will be calculated with Diffusion weighted magnetic resonance imaging gradient b-values of 0 and 1000s/mm2. In the axial ADC map, a region of interest (ROI) will be placed for measurement of ADC values on the renal parenchyma of both kidneys, without any preference for cortex or medulla. Three circular ROIs of size 1 cm2 will be placed-one each at the upper pole, inter-polar region, and lower pole of both kidneys-and 6 total ROIs from bilateral kidneys will be averaged for each patient.

SUMMARY:
Chronic kidney disease (CKD) is a common global public health problem and the average incidence of end-stage renal disease in developing countries is 150 per million population, which is lower than that in the developed world

DETAILED DESCRIPTION:
Since renal parenchymal disease is accompanied by renal dysfunction, monitoring renal function permits assessment of disease progression, and periodic assessment of renal function is necessary for optimal management of a patient with suspected/proven renal disease. Serum creatinine (S Cr), blood urea (BU), and estimated glomerular filtration rate (eGFR) derived from creatinine clearance are useful for monitoring renal function; however, these indirect measures of renal filtration are imperfect and cannot assess single kidney function.

Keeping in view the limitations of serum markers, imaging may play an important role in the evaluation of renal parenchymal disease. Ultrasonography (US) and computed tomographic (CT) scan provide good anatomic images but limited functional information. Although US may show changes in renal echogenicity, it suffers from operator dependency and lacks objectivity. In addition to exposure to ionizing radiation, computed tomography (CT) scan requires use of iodinated contrast material, which is undesirable in patients with renal dysfunction. Magnetic resonance imaging (MRI) has the unique ability to show both structure and function objectively without any radiation exposure to the patient. Functional MRI techniques such as diffusion-weighted imaging (DWI), blood oxygen level-dependent (BOLD) imaging have potential utility in the evaluation of renal function .

ELIGIBILITY:
Inclusion Criteria:

* Patients in different age and sex groups with CKD detected by clinical and laboratory examination.

Exclusion Criteria:

* Patients with any general contraindication to MRI as presence of any paramagnetic substance as pacemakers or in severely ill patients or those with claustrophobia and arrhythmic patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation apparent diffusion coefficient(ADC)of the kidneys for 31 patient with chronic kidney disease by diffusion gradient 0_1000s/mm2 | up to 24hour
  In the axial apparent diffusion coefficient(ADC )map, a region of interest (ROI) will be placed for measurement of ADC values on the renal parenchyma of both kidneys, without any preference for cortex or medulla. Three circular ROIs of size 1 cm2 will be placed-one each at the upper pole, inter-polar region, and lower pole of both kidneys-and 6 total ROIs from bilateral kidneys will be averaged for each patient. The mean ADC values will be recorded for each patient and the relationship of ADC values of different stages of CKD and its relationship with serum markers of renal function will be evaluated.

REFERENCES:
- [Background] Prigent A. Monitoring renal function and limitations of renal function tests. Semin Nucl Med. 2008 Jan;38(1):32-46. doi: 10.1053/j.semnuclmed.2007.09.003. PMID 18096462
- [Background] Squillaci E, Manenti G, Di Stefano F, Miano R, Strigari L, Simonetti G. Diffusion-weighted MR imaging in the evaluation of renal tumours. J Exp Clin Cancer Res. 2004 Mar;23(1):39-45. PMID 15149149